CLINICAL TRIAL: NCT00465491
Title: A Randomized, Controlled Phase III Trial of Picoplatin and BSC Versus BSC Alone in Patients With Small Cell Lung Cancer (SCLC), Refractory or Progressive Within Six Months of Completing First-Line, Platinum-Containing Chemotherapy.
Brief Title: Study of Picoplatin Efficacy After Relapse
Acronym: SPEAR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Poniard Pharmaceuticals (Industry)
Responsible Party: Hazel Breitz, MD, Poniard Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0601
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2009-04-14 (Estimated); Status verified 2009-04

CONDITIONS: Small Cell Lung Cancer
Keywords: refractory; chemotherapy; progressed; second-line treatment; small cell lung cancer; best supportive care; picoplatin
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — amminedichloro(2-methylpyridine)platinum(II)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Picoplatin
  Interventions: Drug: picoplatin
- 2 (Other): BSC
  Interventions: Other: best supportive care

INTERVENTIONS:
Drug: picoplatin — IV picoplatin 150mg/m2 q3wk
  Arms: 1
Other: best supportive care — best supportive care
  Arms: 2

SUMMARY:
Picoplatin is a new type of platinum drug that has been investigated in several clinical trials, and may provide an improved safety profile over current treatment options. This study is designed to compare the efficacy and safety of picoplatin plus Best Supportive Care (BSC) with BSC alone. Best Supportive Care includes care and treatment to optimize the comfort of patients and their ability to function, as well as to minimize the side-effects of anti-cancer treatments.

DETAILED DESCRIPTION:
This Phase 3 study will enroll subjects with Small Cell Lung Cancer (SCLC) who are refractory or progressive within 6 months of completing first-line, platinum-containing chemotherapy. Subjects will be centrally randomized 2:1 to receive picoplatin plus BSC every 3 weeks, or BSC alone. After discontinuation of picoplatin, all subjects will continue to receive BSC and will continue to be evaluated every 3 weeks until discontinuation from the study, death, or the end of the study. After discontinuation of picoplatin, subjects may be treated with another chemotherapy at their physician's discretion and then will be followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of SCLC or combined SCLC/non-small cell lung cancer (NSCLC) defined as SCLC mixed with squamous cell carcinoma, adenocarcinoma, or large cell carcinoma.
* One and only 1 prior cisplatin or carboplatin-containing chemotherapy regimen for SCLC within the scope of the National Comprehensive Cancer Network (NCCN) Guidelines (Section 5.4.1).
* Radiological evidence of SCLC that never responded or progressed within 90 days after completion of first-line therapy (refractory); or responded initially to first-line therapy but progressed between 91 and 180 days after treatment was completed (progressed within 91 to 180 days).
* CT scans of head, chest and abdomen (including adrenal and full extent of liver) with contrast, preferably within 14 days prior to randomization (up to 21 days is allowed if necessary). MRI is acceptable in the case of allergy to contrast agents. The presence or absence of measurable disease gy RECIST must be documented from the baseline CT or MRI scan.
* Patients with brain metastases must have been treated with brain irradiation. Only patients wtih asymptomatic brain metastases are eligible for this study.
* ECOG PS 0, 1 or 2 within 3 days prior to randomization (Appendix II).
* Life expectancy of at least 8 weeks within 3 days prior to randomization.
* At least 21 days must have elapsed since the most recent prior chemotherapy dose, with evidence of hematological recovery.
* At least 14 days must have elapsed since the most recent prior radiotherapy dose.
* At least 14 days must have elapsed since prior surgery except for the placement of venous access device or bronchoscopy.
* Subject must be recovered to ≤ Grade 1 toxicity from all non-hematological adverse effects of prior therapies (excluding alopecia).
* Age 18 years or over.
* ANC ≥ 1.5 x 109/L.
* Platelet count ≥ 100 x 109/L.
* Hemoglobin of ≥ 90 g/L (transfusion permitted to achieve this hemoglobin).
* Aspartate aminotransferase, alanine aminotransferase, and lactate dehydrogenase levels ≤ 2.5 times upper limit of normal (ULN) or ≤ 5 times ULN if liver involvement is present.
* Bilirubin of ≤ 1.5 times upper limit of normal (ULN).
* Blood urea nitrogen ≤ 1.5 times ULN (hypovolemic subjects may be hydrated to achieve this BUN).
* Creatinine clearance of ≥ 50 mL/min, as calculated by the Cockcroft-Gault formula (Appendix III).
* Women of childbearing potential must have a negative pregnancy test (serum or urine). Sexually active couples of child-bearing potential must agree to use appropriate birth control methods during chemotherapy and for 3 months after chemotherapy.
* Signed informed consent.

Exclusion Criteria:

* Prior radiotherapy that included ≥ 30% of the bone marrow (Appendix IV).
* Pleural effusion as the only radiological evidence of SCLC.
* Untreated or symptomatic brain or central nervous system (CNS) metastases.
* Grade 2 or higher peripheral neuropathy.
* Significant cardiac disease, defined as myocardial infarction within 3 months prior to randomization, congestive heart failure classified by the New York Heart Association as Class III or IV (Appendix V), uncontrolled cardiac arrhythmias, poorly controlled or unstable angina, or electrocardiographic evidence of acute ischemia.
* Serious medical or psychiatric illness that could potentially interfere with the completion of study treatment according to this protocol, e.g., active infection, Crohn's disease, ulcerative colitis, etc.
* Use of other investigational drugs within 30 days prior to randomization.
* Breast-feeding.
* History of any other malignancy within 5 years, with the exception of treated non-melanoma skin cancer or carcinoma in situ of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
overall survival | death

SECONDARY OUTCOMES:
objective response rate | progression
disease control rate | progression
duration of response | progression
progression-free survival | death

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Hazel Breitz, M.D., Study Director — Poniard Pharmaceuticals
Locations (143):
- Argentina (11):
  - Consultorios Privados, Buenos Aires
  - Clinica Constituyentes, Buenos Aires
  - CETEN Centro de Estudio y Tratamiento de Enfermedades Neoplasicas, Buenos Aires
  - IADT (Insttituto Argentino de Diagnostico y Tratamiento S.A.), Buenos Aires
  - Centro Oncologico, Buenos Aires
  - Instituto Alexander Fleming, Buenos Aires
  - PALIAR, Buenos Aires
  - IONC, Córdoba
  - Centro Medico San Roque, San Miguel de Tucumán
  - Centro Oncologico de Rosario, Santa Fe
  - ISIS Clinica Especializada, Santa Fe
- Belarus (5):
  - Institution of Healthcare "Grodno Regional Clinical Hospital, Grodno
  - Gomel Regional Oncological Dispensary, Homyel
  - Minsk City Clinical Oncology Dispensary, Minsk
  - Research Institute of Oncology and Medical Radiology named by N.N. Aleksandrov, Minsk
  - Vitebsk Regional Oncology Dispensary, Vitebsk
- Bosnia and Herzegovina (2):
  - Clinic for Lung Diseases, Clinical Center, Banja Luka, Banja Luka
  - Clinic of Pulmonary Diseases Podhrastovi, Sarajevo
- Bulgaria (8):
  - Multiprofile Hospital for Active Treatment, Dr. Tota Venkova, Gabrovo
  - University Multifunctional Hospital for Active Treatment "Dr. Georgi Stranski", Pleven
  - District Dispensary for Cancer Diseases with Inpatient Hospital Plovdiv, Plovdiv
  - Regional Oncodispensary with Inpatient Sector, Rousse
  - Inter-district Dispensary for Cancer Diseases w/Inpatient Hospital, Shumen
  - Regional Oncodispensary with Inpatient Sector-Sofia District, Sofia
  - Inter-district Dispensary for Cancer Disease w/Inpatient Hospital "Dr. Marko Markov", Varna, Varna
  - Multiprofile Hospital for Active Treatment "St. Marina", Varna
- Instituto Nacional de Cancer, Santiago, Chile
- Croatia (4):
  - Clinical Hospital, Dubrovnik
  - Clinical Hospital, Osijek
  - Clinical Hospital Split, Split
  - Clinic for Pulmonary Diseses "Jordanovac", Zagreb
- Hungary (3):
  - St. George County Hospital, Fejer County
  - University of Szeged, Szeged
  - General Rehablitation and Medicinal Bath Hospital, Szombathely
- India (24):
  - Gujrat Cancer Research Institute, Asarwa, Ahmadabad
  - Kidwai Memorial Institute of Oncology, Bangalore, Karnataka
  - Lakeshore Hospital and Research Center, Kochi, Kerala
  - Shatabdi Superspeciality Hospital, Nashik, Maharashtra
  - Curie Centre of Oncology, Bangalore
  - Jawaharlal Nehru Cancer Hospital and Research Centre, Bhopal
  - Apollo Speciality Hospital, Chennai
  - MNJ Institute of Oncology, Hyderabaad
  - Indo American Institute of Oncology, Hyderabaad
  - Yashoda Group of Hospitals, Hyderabad
  - SEAROC Cancer Center, Jaipur
  - Institute of Post Graduate Medical Education and Research, Kolkata
  - Orchid Nursing Home, Kolkata
  - King George Medical University, Lucknow
  - KMC (Karturba Medical College) Hospital, Manipal
  - Jaslok Hospital and Research Centre, Mumbai
  - Tata Memorial Centre, Mumbai
  - Sir Ganga Ram Hospital, New Delhi
  - Rajiv Gandhi Cancer Institute, Delhi, New Delhi
  - Mahaveer Cancer Sansthan, Patna
  - Jahangir Hospital and Research Centre, Pune
  - Smt. Vasantben R. Desai Cancer Research Center, Rajkot
  - Regional Cancer Centre, Trivandrum
  - King George Hospital, Visakhapatnam
- Latvia (2):
  - Daugavas Hospital, Daugavpils
  - Paul Stradins Clincial University Hospital, Riga
- Special Hospital for Pulmonary Diseases, Nikšić, Montenegro
- Poland (13):
  - Silesian Medical University in Katowice, Zabrze, Dolny Slask
  - Dolnoslaskie Centre of Lung Diseases, Wroclaw, Lower Silesian Voivodeship
  - Kujawsko-Pomorski Centre of Pulmonology, Bydgoszcz
  - NMP, Memorial Voyvodship Hospital, Częstochowa
  - Dr. Bieganski Memorial Regional Specialsitic Hospital, Grudziądz
  - Regional Hospital, Department of Pulmonary Diseases and Chemotherapy, Krakow
  - Independent Public Group for Tuberculosis and Lung Disease in Olsztyn, Olsztyn
  - Department of Clinical Oncology, Wielkopolskie Centre of Lung Diseases and Tuberculosis, Poznan
  - Conservative Outpatient Oncology Department, Voyevodship Hospital in Plock, Płock
  - Department of Pulmonology, Voyvodship Specialsitic Hospital in Radom, Radom
  - SP ZOZ Voyevodship Specialistic Hospital #3, Rybnik
  - Department of Chemotherapy, Prof. A. Sokolowski Memorial Specialistic Hospital in Szczecin, Szczecin
  - Department of Clinical Oncology, SP ZOZ, Yoyvodship Specialistic Hospital, Torun
- Romania (11):
  - Prof. Dr. Ion Chiricuta, Institute of Oncology Cluj-Napoca, Cluj-Napoca, Cluj
  - Baia Mare "Constantin Opris" County Emergency Hospital, Baia Mare, Maramureş
  - IANULI Medconsult SRL, Bucharest
  - Bucharest Institute of Oncology, Bucharest
  - Prof. Dr. Ion Chircuta, Oncology Institute, Cluj-Napoca
  - Clinical Emergency County Hospital Constanta, Constanța
  - Medical Oncology Center Iasi, Iași
  - Schuller Municipal Hospital Ploiesti-Medical Oncology Department, Ploieşti
  - Clinical County Hospital, Sibiu
  - Sf. loan cel Nou, Emergency County Hospital, Suceava
  - OncoMed, Timișoara
- Russia (51):
  - Buryatia Republican Oncology Center, Ulan-Ude, Buryatiya Republic
  - Regional Oncology Center, Birobidzhan, Jewish Republic
  - Republican Oncology Center of the Ministry of Healthcare of Karelia Republic, Petrozavodsk, Karelia Republic
  - Komi Republican Oncology Center, Syktyvkar, Komi
  - Clinical Oncology Center, Kazan', Tatarstan Republic
  - Kazan Oncology Center, Kazan', Tatarstan Republic
  - Arkhangelsk Regional Clinical Oncology Center, Arkhangelsk
  - Altai Regional Oncology Center, Barnaul
  - Chelyabinsk Regional Oncology Center, Chelyabinsk
  - City Hospital #1, Cherepovets
  - Chita Regional Oncology Center, Chita
  - Regional Oncology Center, Engel's
  - Regional Oncology Center, Irkutsk
  - Ivanovo Regional Oncology Center, Ivanovo
  - Republican Clinical Oncology Center of the Republic of Udmurtia, Izhevsk
  - Kaluga Regional Oncology Center, Kaluga
  - Regional Clinical Oncology Center, Khabarovsk
  - Regional Clinical Oncology Center, Kirov
  - City Oncology Center, Komsomolsk-on-Amur
  - Krasnodar Clinical Oncology, Krasnodar
  - Regional Clinical Hospital #1, Krasnodar
  - Kurst Regional Oncology Center, Kurst
  - Lipetsk Regional Oncology Center, Lipetsk
  - Magnitogorsk Clinical Oncology Hospital, Magnitogorsk
  - Blokhin Russian Oncology Research Center, Moscow
  - Central Clinical Hospital and Outpatient Unit of the Medical Center under the Russian Presidential Administration, Moscow
  - Semashko Central Clinical Hospital #2 under Russian Railways, Moscow
  - Novorossiysk Oncology Center, Novorossiysk
  - City Clinical Hospital #1, Novosibirsk
  - Medical Radiology Research Center under RAMS, Obnninsk
  - Orenburg Regional Clinical Oncology Center, Orenburg
  - Orel Oncology Center, Oryol
  - Regional Oncology Center, Penza
  - Pyatigorsk Affiliate of Stavropol Regional Clinical Oncology Center, Pyatigorsk
  - St. Petersburg City Multifield Hospital #2, Saint Petersburg
  - St. Petersburg Pavlov State Medical University, Saint Petersburg
  - Pavlov St. Petersburg State Medical University, Pulmonology Research Institute, Saint Petersburg
  - City Clinical Oncology Center, Thoracic Oncology Department #6, Saint Petersburg
  - Ogarev Mordovian State University, Saransk
  - State Higher Education Institution Saratov State Medical University under the Federal Agency for Healthcare and Social Development, Saratov
  - Oncology Center, Sochi
  - Tambov Regional Oncology Center, Tambov
  - Tomsk Regional Oncology Center, Tomsk
  - Tula Regional Oncology Center, Tula
  - Ufa, Republican Oncology Center, Ufa
  - Primorsky Regional Oncology Center, Vladivostok
  - Volgograd Regional Clinical Oncology Center#1, Volograd
  - Voronezh Regional Clinical Oncology Center, Voronezh
  - Regional Clinical Oncology Hospital, Yaroslavl
  - Sverdlovsk Regional Oncology Center, Yekaterinburg
  - Republican of Clinical Hospital, Mariy-El Republican, Yoshkar-Ola
- Serbia (2):
  - Clinic for Pulmonary Diseases and TBC, Knez-Selo
  - Institute for Pulmonary Diseases of Vijvodina, Vijvodina
- Ukraine (5):
  - Volyn Regional Oncology Center, Lutsk
  - Public Treatment and Prevention Institution Mariupol City Interdistrict Oncology Center, Mariupol
  - Sumy Regional Oncology Center, Sumy
  - Ternopol Regional Clinical Oncology Center, Ternopil
  - Zaporozhye Regional Clinical Oncology Center, Zaporizhzhya

REFERENCES:
- [Background] Raynaud FI, Boxall FE, Goddard PM, Valenti M, Jones M, Murrer BA, Abrams M, Kelland LR. cis-Amminedichloro(2-methylpyridine) platinum(II) (AMD473), a novel sterically hindered platinum complex: in vivo activity, toxicology, and pharmacokinetics in mice. Clin Cancer Res. 1997 Nov;3(11):2063-74. PMID 9815598
- [Background] Beale P, Judson I, O'Donnell A, Trigo J, Rees C, Raynaud F, Turner A, Simmons L, Etterley L. A Phase I clinical and pharmacological study of cis-diamminedichloro(2-methylpyridine) platinum II (AMD473). Br J Cancer. 2003 Apr 7;88(7):1128-34. doi: 10.1038/sj.bjc.6600854. PMID 12671715
- [Background] Giaccone G, O'Brien ME, Byrne MJ, Bard M, Kaukel E, Smit B. Phase II trial of ZD0473 as second-line therapy in mesothelioma. Eur J Cancer. 2002 Dec;38 Suppl 8:S19-24. doi: 10.1016/s0959-8049(02)80018-1. PMID 12647701
- [Background] Treat J, Schiller J, Quoix E, Mauer A, Edelman M, Modiano M, Bonomi P, Ramlau R, Lemarie E. ZD0473 treatment in lung cancer: an overview of the clinical trial results. Eur J Cancer. 2002 Dec;38 Suppl 8:S13-8. doi: 10.1016/s0959-8049(02)80016-8. PMID 12645908
- [Background] Gore ME, Atkinson RJ, Thomas H, Cure H, Rischin D, Beale P, Bougnoux P, Dirix L, Smit WM. Results of ZD0473 in platinum-pretreated ovarian cancer: analysis according to platinum free interval. Eur J Cancer. 2002 Dec;38 Suppl 8:S7-12. doi: 10.1016/s0959-8049(02)80014-4. PMID 12645907
- [Background] Holford J, Raynaud F, Murrer BA, Grimaldi K, Hartley JA, Abrams M, Kelland LR. Chemical, biochemical and pharmacological activity of the novel sterically hindered platinum co-ordination complex, cis-[amminedichloro(2-methylpyridine)] platinum(II) (AMD473). Anticancer Drug Des. 1998 Jan;13(1):1-18. PMID 9474239
- [Background] Holford J, Sharp SY, Murrer BA, Abrams M, Kelland LR. In vitro circumvention of cisplatin resistance by the novel sterically hindered platinum complex AMD473. Br J Cancer. 1998;77(3):366-73. doi: 10.1038/bjc.1998.59. PMID 9472630
- [Background] Rogers P, Boxall FE, Allott CP, Stephens TC, Kelland LR. Sequence-dependent synergism between the new generation platinum agent ZD0473 and paclitaxel in cisplatin-sensitive and -resistant human ovarian carcinoma cell lines. Eur J Cancer. 2002 Aug;38(12):1653-60. doi: 10.1016/s0959-8049(02)00107-7. PMID 12142057
- [Background] Sharp SY, O'Neill CF, Rogers P, Boxall FE, Kelland LR. Retention of activity by the new generation platinum agent AMD0473 in four human tumour cell lines possessing acquired resistance to oxaliplatin. Eur J Cancer. 2002 Nov;38(17):2309-15. doi: 10.1016/s0959-8049(02)00244-7. PMID 12441268
- [Background] Kawamura-Akiyama Y, Kusaba H, Kanzawa F, Tamura T, Saijo N, Nishio K. Non-cross resistance of ZD0473 in acquired cisplatin-resistant lung cancer cell lines. Lung Cancer. 2002 Oct;38(1):43-50. doi: 10.1016/s0169-5002(02)00175-7. PMID 12367792
- See also: Poniard Pharmaceuticals, Inc. — http://www.poniard.com